CLINICAL TRIAL: NCT03793855
Title: Effectiveness of a Nutritional Strategy for Glycemic Control in Patients With Type 2 Diabetes Mellitus Users of a Public Health System: NUGLIC Study
Brief Title: Nutritional Strategy for Glycemic Control in Patients With Type 2 Diabetes Mellitus (NUGLIC)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital do Coracao (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NUGLIC
Record Dates: First submitted 2019-01-03; First posted 2019-01-04 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2022-02

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutritional Strategy (Experimental): Nutritional counseling based on the quality of the diet, the Food Guide for the Brazilian Population and concepts of mindfulness and mindful eating; dietary guidance based on feasible goals built together (patient and nutritionist).
  Interventions: Behavioral: Nutritional Strategy
- Dietary Prescription (Active Comparator): Individualized dietary prescription according to the guidelines of the Brazilian Society of Diabetes.
  Interventions: Behavioral: Dietary Prescription

INTERVENTIONS:
Behavioral: Nutritional Strategy — Counseling based on dietary goals and mindfulness techniques.
  Arms: Nutritional Strategy
Behavioral: Dietary Prescription — Dietary prescription according to guidelines.
  Arms: Dietary Prescription

SUMMARY:
Adherence to a healthy dietary pattern is part of the self-care of patients with type 2 diabetes mellitus (T2DM), and may contribute substantially to therapeutic target goals and to a better quality of life as well. However, not all nutritional recommendations aimed at these patients are easily applicable in clinical practice. The primary objective of the study is to evaluate the effectiveness of a nutritional strategy for glycemic control in patients with T2DM users of a Public Health System after 6 months of follow-up. As secondary objectives, we will evaluate the impact of the proposed strategy on self-care and on the quality of life of the patients. In this randomized multicenter open-label randomized trial, 370 patients >30 years old with T2DM, glycated hemoglobin (HbA1C) ≥7% at the moment of the screening and who have not received or received nutritional counseling for at least 06 months will be enrolled. Patients allocated to the control group will receive individualized dietary prescription according to the guidelines of the Brazilian Society of Diabetes. Nutritional counseling in the intervention group will be performed based on the quality of the diet, the Food Guide for the Brazilian Population and concepts of mindfulness and mindful eating; all dietary guidance will be based on feasible goals built together (patient and nutritionist), and no diet will be prescribed for intervention group. In both groups, patients will receive glymeters for residential self-monitoring of glycemic levels. On-site follow-up visits will be carried out at 30, 60, 90, and 180 days (final consultation). At 120 and 150 days, participants in the intervention group will receive motivational messages via e-mail or SMS (for these patients, consultation of 30 days will be a group meeting). Laboratory tests (lipid and glycemic profile, serum creatinine, serum sodium, urinary sodium, serum potassium, urinary potassium and albuminuria) will be performed at baseline and 180 days; anthropometric indexes and blood pressure will be also evaluated.

ELIGIBILITY:
Inclusion Criteria: >30 years old with medical diagnosis of T2DM, glycated hemoglobin (HbA1C) ≥7% at the moment of the screening and who have not received or received nutritional counseling for at least 06 months.

Exclusion Criteria:

* Patients with type 1 DM (T1DM), latent autoimmune diabetes in adults (LADA) or HbA1C ≥ 12%;
* Severe neuropathy;
* Chronic kidney disease;
* Active cancer or life expectancy <6 months;
* Chemical dependence or use of antipsychotic drugs;
* Autoimmune disease or chronic use of steroids;
* Gastroparesis;
* Pregnancy, lactation, gestational DM;
* Acute coronary syndrome (ACS) in the last 60 days;
* Wheelchair users;
* Extreme obesity (body mass index [BMI] ≥40kg/m²);
* Cognitive, neurological or psychiatric condition that prevents participation in the study;
* Participation in other clinical trials.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370 (Actual)
Dates: Start 2019-05-06 (Actual); Primary Completion 2021-09-28 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
HbA1C | 6 months
  Glycated hemoglobin, in %
GC | 6 months
  Glycemic control, defined as either having HbA1C > 7% at baseline and achieving HbA1C ≤ 7% after follow-up or having HbA1C < 7% at baseline and reducing anti-diabetic drugs after follow-up.

SECONDARY OUTCOMES:
FG | 6 months
  Fasting glucose, in mg/dL
SBP | 6 months
  Systolic blood pressure, in mmHg
DBP | 6 months
  Diastolic blood pressure, in mmHg
HDL-c | 6 months
  HDL cholesterol, in mg/dL
LDL-c | 6 months
  LDL cholesterol, in mg/dL; it will be obtained by the Martin´s mathematical formula
TC | 6 months
  Total cholesterol, in md/dL
TG | 6 months
  Serum triglycerides, in mg/dL
Castelli Index I | 6 months
  Castelli Index I, obtained by the mathematical formula TC/HDL-c
VLDL-c | 6 months
  VLDL cholesterol, in mg/dL; it will be obtained by the mathematical formula TG/5
NHDL | 6 months
  Non-HDL cholesterol, in mg/dL; it will be obtained by the mathematical formula TC - HDL-c
Castelli Index II | 6 months
  Castelli Index II, obtained by the mathematical formula LDL-c/HDL-c
BW | 6 months
  Body weight, in kg
WC | 6 months
  Waist circumference, in cm
BMI | 6 months
  Body mass index, in kg/m2; it will be obtained by the mathematical formula (BW/height*height)
Cr | 6 months
  Creatinine, in mg/dL
GFR | 6 months
  Glomerular filtration rate, in ml/min/1.73m2
Sodium (s) | 6 months
  Serum sodium, in mEq/L
Sodium (u) | 6 months
  Urinary sodium, in mEq/L
Potassium (s) | 6 months
  Serum potassium, in mEq/L
Potassium (u) | 6 months
  Urinary potassium, in mEq/L
ALB | 6 months
  Albuminuria, in mg/g
B-PAID | 6 months
  Quality of life evaluated by the Brazilian version of the Problem Areas in Diabetes Scale. The scale consists of 20 questions; it uses a score from 0 to 100, in which the maximum score is configured as greater suffering. The possible response options are divided on a 5-point Likert scale, ranging from: "Not a problem=0", "Small problem=1", "Moderate problem=2", "Almost serious problem=3", "Serious problem=4". A cut-off point equal or greater 40 indicates a high degree of emotional distress.
DSCA | 6 months
  Self-care evaluated by the Brazilian version of the Diabetes Self-Care Activities. The questionnaire has six domains and 15 items for assessment of the diabetes self-care; it is based on the number of days per week in which the respondent has a given behavior, with each item scoring from 0 to 7 points (i.e. 0 is the least desirable situation and 7 is the most desirable one). At least five days for each self-care activity is considered adequate.
DQ | 6 months
  Diet quality, evaluated by the modified Alternative Healthy Eating Index (mAHEI)

OTHER OUTCOMES:
TT | 6 months
  Therapeutic targets, defined as the proportion of participants who reached the following therapeutic targets: SBP/DBP < 130/80 mmHg; HbA1C <7%; LDL-c <100 mg/dL; BMI < 25 kg/m2 or weight loss > 7%
ADD | 6 months
  Anti-diabetic drugs, defined as the type and proportion of anti-diabetic drugs used

CONTACTS AND LOCATIONS:
Overall Officials: Aline Marcadenti, PhD, Principal Investigator — Hospital do Coracao
Locations (8):
- Brazil (8):
  - Universidade Federal de Juiz de Fora, Governador Valadares
  - Universidade Federal de Lavras, Lavras
  - Hospital de Clínicas de Porto Alegre - Universidade Federal do Rio Grande do Sul, Porto Alegre
  - Universidade Federal de Ciências da Saúde de Porto Alegre, Porto Alegre
  - Instituto Estadual de Cardiologia Aloysio de Castro, Rio de Janeiro
  - Universidade Federal da Bahia, Salvador
  - Hospital do Coracao, São Paulo
  - Universidade Federal de Viçosa, Viçosa

IPD SHARING:
Plan to Share IPD: Yes
Data and materials will be available upon reasonable request for the corresponding author, after filling a specific form provided by IP-HCor and considering institutional data sharing politics.
Time Frame: Data will be available after main paper publication.